CLINICAL TRIAL: NCT05348915
Title: An Open-label Extension Study to Evaluate the Long-term Safety of Inclacumab Administered to Participants With Sickle Cell Disease Who Have Participated in an Inclacumab Clinical Trial
Brief Title: A Study to Evaluate the Long-term Safety of Inclacumab Administered to Participants With Sickle Cell Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to terminate study based on results of parent study GBT2104-131.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT2104-133; 2020-005289-32 (EudraCT Number); C5361003 (Other: Alias Study Number)
Record Dates: First submitted 2022-03-29; First posted 2022-04-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis; Vaso-occlusive Pain Episode in Sickle Cell Disease
Keywords: blood disorders; hemoglobin; red blood cells; RBCs; sickle-like shape; mutation in hemoglobin gene; Sickle Cell Disease; SCD; Vaso-occlusive Crisis; VOC; SCA; Open Label
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Hematologic Diseases | interventions — inclacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inclacumab 30 mg/kg (Experimental): Inclacumab 30 mg/kg administered intravenously (IV)
  Interventions: Drug: Inclacumab

INTERVENTIONS:
Drug: Inclacumab — Inclacumab will be supplied in single use 10 mL vials at a concentration of 50 mg/mL. One vial contains 500 mg of inclacumab. This is a liquid concentrate for IV infusion.

SUMMARY:
This study is an open-label study to evaluate the safety of long-term administration of inclacumab in participants with sickle cell disease (SCD). Participants in this study will have completed a prior study of inclacumab.

DETAILED DESCRIPTION:
The study will include approximately 520 adult and adolescent participants (≥ 12 years of age) with SCD.

All participants will receive inclacumab 30 mg/kg administered intravenously every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all the following criteria will be eligible for study enrollment:

1. Male or female participant with SCD who participated and received study drug in a GBT-Sponsored inclacumab clinical study.
2. Participant has completed the originating inclacumab study within 30 calendar days of the Day 1 Visit. Participants who discontinued study drug in the originating study due to a non-study drug-related AE, but who remained on study, may be eligible for treatment in this study provided the AE does not pose a risk for treatment with inclacumab.
3. Female participants of childbearing potential are required to have a negative urine pregnancy test prior to dosing on Day 1.

   Note: Female participants who become of childbearing potential during the study must be willing to have a negative urine pregnancy test to remain in the study.
4. If sexually active, female participants of childbearing potential must consistently use highly effective methods of contraception consistently throughout the study and for at least 165 days after the last dose of study drug. If sexually active, male participants must use barrier methods of contraception until 165 days after the last dose of study drug.
5. Participant has provided written informed consent/assent. For underage participants, both the consent of the participant's legal representative or legal guardian and the participant's assent (where applicable) must be obtained based on local requirement.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria will not be eligible for study enrollment:

1. Female participant who is breastfeeding or pregnant.
2. Participant had an infusions-related reaction (IRR) in the originating inclacumab clinical study.
3. Participant withdrew consent from the originating inclacumab clinical study.
4. Participant was lost to follow-up from the originating inclacumab clinical study.
5. Participant has any medical, psychological, safety, or behavioral conditions that, in the opinion of the Investigator, may confound safety interpretation, interfere with compliance, or preclude informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs). | Day 1 through study completion, an estimate of 5 years

SECONDARY OUTCOMES:
Annualized rate of VOCs | Day 1 through study completion, an estimate of 5 years
Annualized rate of VOCs that require admission to a healthcare facility and treatment. | Day 1 through study completion, an estimate of 5 years
Annualized number of days of inpatient hospitalization for a VOC. | Day 1 through study completion, an estimate of 5 years
Annualized rate of all SCD-related urgent care visits to the clinic, emergency room, and hospital. | Day 1 through study completion, an estimate of 5 years
Proportion of total days missed from school or work due to SCD pain symptoms for the first 48 weeks. | Day 1 through study completion, an estimate of 5 years
Annualized rate of complicated VOCs. | Day 1 through study completion, an estimate of 5 years
Annualized rate of RBC transfusions. | Day 1 through study completion, an estimate of 5 years

OTHER OUTCOMES:
Plasma pharmacokinetic (PK) of inclacumab as assessed by population PK analysis using nonlinear mixed-effects modeling. | Day 1 through Week 48
  Inclacumab concentrations will be measured from plasma samples. Population PK analysis using nonlinear mixed effects modeling will be performed to characterize inclacumab PK in plasma.
Incidence of anti-drug antibodies (ADA) to inclacumab. | Day 1 through Week 48
PD parameter (P-selectin inhibition) | Day 1 through Week 48
PD parameter (Platelet Leukocyte Aggregation) | Day 1 through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (18):
  - Strada Patient Care Center, Pediatric Hematology, Mobile, Alabama
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - South Alabama Medical Science Foundation, Mobile, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC Irvine Medical Center, Orange, California
  - UConn-Neag Comprehensive Cancer Center, Farmington, Connecticut
  - University of Illinois at Chicago (UIC) Clinical Research Center, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System (UI Health), Chicago, Illinois
  - Brigham And Woman's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute IDS Pharmacy, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospitals - Michigan Medicine, Ann Arbor, Michigan
  - Jacobi Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - DUMC Investigational Drug Services Pharmacy, Durham, North Carolina
  - McGovern Medical School at UTHealth, Houston, Texas
  - UT Health Science Center at Houston - Clinical Research Unit at Memorial Hermann Hospital, Houston, Texas
  - UT Physicians Comprehensive Sickle Cell Center Houston, Houston, Texas
- Brazil (9):
  - Instituto D'Or de Pesquisa e Ensino - Hospital São Rafael, Salvador, Estado de Bahia
  - Multihemo Servicos Medicos S/A, Recife, Pernambuco
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto Estadual de Hematologia Arthur Siqueira Cavalcanti - HEMORIO, Rio de Janeiro
  - Hospital Samaritano Higienópolis/Esho Empresa De Servicos Hospitalares S.A, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo
  - CEPEC-Centro de Pesquisa Clinica, São Paulo
- Colombia (2):
  - Clinica de la Costa Ltda., Barranquilla, Atlántico
  - Sociedad de Oncología y hematología del Cesar, Valledupar, Cesar Department
- Kenya (5):
  - KEMRI/CRDR Siaya Clinical Research Annex, Kisumu, Siaya County
  - International Cancer Institute, Eldoret
  - Gertrude's Children's Hospital, Nairobi
  - Kenya Medical Research Institute - Centre for Respiratory Disease Research, Nairobi
  - Strathmore University CREATES, Nairobi
- Lebanon (2):
  - American University of Beirut Medical Center, Hamra, Beyrouth
  - Nini Hospital, Tripoli, North Lebanon
- Nigeria (8):
  - University of Calabar Teaching Hospital, Calabar, Cross River State
  - National Hospital Abuja, Abuja, Federal Capital Territory
  - University of Abuja Teaching Hospital, Gwagwalada, Federal Capital Territory
  - Ahmadu Bello University Teaching Hospital, Zaria, Kaduna State
  - University of Nigeria Teaching Hospital, Enugu
  - Barau Dikko Teaching Hospital/Kaduna State University, Kaduna
  - Aminu Kano Teaching Hospital, Kano
  - Department of Pediatrics, College of Medicine, Lagos University Teaching Hospital, Lagos
- Sultan Qaboos University Hospital, Muscat, Oman
- Prince Mohammed bin Nasser Hospital, Jizan, Southern, Saudi Arabia
- National Institute for Medical Research (NIMR), Dar es Salaam, Tanzania
- Turkey (Türkiye) (3):
  - Acibadem Adana Hastanesi Cocuk Hematoloji Onkoloji, Adana
  - Baskent University Adana Appl. and Research Central, Yuregir Baskent Hospital Hematology, Adana
  - Hacettepe University Ihsan Dogramaci Children Hospital, Ankara

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT2104-133